CLINICAL TRIAL: NCT04029415
Title: The Study of the Antimicrobial Resistance of Helicobacter Pylori in Shandong Province
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2018SDU-QILU-G114
Record Dates: First submitted 2019-07-21; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Helicobacter Pylori
Keywords: antimicrobial resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The gastric mucosa of the lesser curvature of gastric antrum and the greater curvature of the stomach
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The antimicrobial resistance of helicobacter pylori in Shandong province was analyzed by helicobacter pylori antibiotic sensitivity test.And the map of antimicrobial resistance of helicobacter pylori was constructed to provide clinical guidance for selecting effective eradication program and improve the eradication rate.

DETAILED DESCRIPTION:
The patients with positive H. pylori infection that was not eradicated by previous therapies will accept the gastroscopy. The mucosa of the lesser curvature of gastric antrum and the greater curvature of the stomach will progress helicobacter pylori antibiotic sensitivity test to detect the antimicrobial resistance of helicobacter pylori.The antimicrobial resistance of helicobacter pylori in Shandong province will be described by frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18 and 70 years old, with positive H. pylori infection that was not eradicated by previous therapies are included. The H. pylori infection is confirmed by the positive rapid urease test or 13C-breath test.

Exclusion Criteria:

* Patients with significant underlying disease including liver, cardiac, pulmonary, and renal diseases, neoplasia, coagulopathy and genetic diseases, history of gastric surgery, pregnancy, breast-feeding, active gastrointestinal bleeding, the use of PPI, NSAID or antibiotics during the 4 weeks prior to enrolment, and previous history of allergic reactions to any of the medications used in this protocol. Patients previously treated with H. pylori eradication regimens or those unwilling to participate in the study were also excluded.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The patients in Shandong province, aged between 18 and 70 years old, with positive H. pylori infection that was not eradicated by previous therapies are included.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial resistance rate | 3years
  The antimicrobial resistance rate will be described by the frequency and percentage.

SECONDARY OUTCOMES:
The influence factors of the antimicrobial resistance rate | 3years
  The chi-square test will be used to compare the influence factors of the antimicrobial resistance rate.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Study Chair — Qilu Hospital of Shandong University; Tian Ma, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China